CLINICAL TRIAL: NCT00331500
Title: A Comparative Study of Olopatadine 0.2% Versus Vehicle in Patients With Seasonal Allergic Conjunctivitis or Rhinoconjunctivitis
Brief Title: Olopatadine 0.2% for the Treatment of Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-04-60
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2008-06

CONDITIONS: Allergic Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Olopatadine Hydrochloride 0.2% (Experimental): Olopatadine hydrochloride ophthalmic solution, 0.2%, 1 drop in each eye, once-daily in the morning for 6 weeks
  Interventions: Drug: Olopatadine Hydrochloride Ophthalmic Solution, 0.2%
- Vehicle (Placebo Comparator): Olopatadine hydrochloride ophthalmic solution vehicle, 1 drop in each eye, once-daily in the morning for 6 weeks
  Interventions: Drug: Olopatadine Hydrochloride Ophthalmic Solution Vehicle

INTERVENTIONS:
Drug: Olopatadine Hydrochloride Ophthalmic Solution, 0.2%
  Arms: Olopatadine Hydrochloride 0.2%
Drug: Olopatadine Hydrochloride Ophthalmic Solution Vehicle — Inactive ingredients used as a placebo comparator
  Arms: Vehicle

SUMMARY:
The purpose of this study is to demonstrate that Olopatadine 0.2% is superior to vehicle in the treatment of the signs and symptoms associated with allergic conjunctivitis or rhinoconjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* History of seasonal allergic conjunctivitis or rhinoconjunctivitis, a positive grass antigen challenge reaction (skin test), and a positive response to grass in the Conjunctival Allergen Challenge (CAC) model

Exclusion Criteria:

* Under 10 years of age

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2006-04-18 (Actual); Primary Completion 2006-07-27 (Actual); Study Completion 2006-07-27 (Actual)

PRIMARY OUTCOMES:
Daily ocular itching and redness scores | Up to Day 14

SECONDARY OUTCOMES:
Percentage of patients with daily ocular itching and redness scores of 0 | Up to Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Alcon, A Novartis Company, Study Director — Alcon, a Novartis Company

REFERENCES:
- [Result] https://www.ncbi.nlm.nih.gov/pubmed/23379201